CLINICAL TRIAL: NCT02144064
Title: Pregnancy Outcomes in Women With Unexplained Recurrent Pregnancy Loss Treated With Low Dose Aspirin and Unfractionated Heparin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, khalid abd aziz mohamed, lecturer of ob/gyn, Benha University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: khalid-ahmed 3
Record Dates: First submitted 2014-05-16; First posted 2014-05-21 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Recurrent Pregnancy Loss
Keywords: Aspirin, heparin, pregnancy, recurrent pregnancy loss
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A(heparin group) (Active Comparator): Group A (n = 100) are put on Inj. UFH (Cal-heparin) 5000 U subcutaneous twice daily plusAspirin 81 mg/day (Juspirin) with the ﬁrst positive pregnancy test, Inj. UFH is given either into anterior abdominal wall or anterior aspect of thigh subcutaneously
  Interventions: Drug: Heparin
- Group B (No Intervention): group B (n = 100) receive no thing

INTERVENTIONS:
Drug: Heparin — Group A (n = 100) are put on Inj. UFH (Cal-heparin) 5000 U subcutaneous twice daily plusAspirin 81 mg/day (Juspirin) with the ﬁrst positive pregnancy test, Inj. UFH is given either into anterior abdominal wall or anterior aspect of thigh subcutaneously
  Other Names: cal-heparin 5000 U; juspirin
  Arms: Group A(heparin group)

SUMMARY:
Objective To determine maternal and fetal outcomes in women with Unexplained RPL managed with aspirin or unfractionated heparin (UFH) plus aspirin during pregnancy.

Design: prospective clinical controlled study. Setting: high-risk pregnancy unit- Benha university hospital. Methods: Pregnant women with unexplained recurrent miscarriage attending high-risk pregnancy unit. 200 selected patients with previous unexplained recurrent miscarriage are divided into 2 groups: group A (n = 100) receive low-dose aspirin (81 mg once daily orally) plus heparin (5000 IU) every 12 h with the ﬁrst positive pregnancy test while group B (n = 100) receive no thing .

Main outcome measures: Maternal outcomes included thromboembolic and haemorrhagic complications and pregnancy-induced hypertension .Prematurity, intrauterine growth restriction and neonatal death were considered as maternal and fetal complications

DETAILED DESCRIPTION:
This prospective comparative, controlled clinical study is conducted at Department of Obstetrics and Gynecology, Benha University Hospital, and a private center, from June 2012 . After approval of the study protocol by the Local Ethical Committee and obtaining written fully informed patients' consents. All patients are interviewed about their medical, personal, family, obstetrical and thrombosis history. All patients included in study complain of three or more unexplained consecutive spontaneous abortions.

All patients (n=200) are in good general health without previous history of Diabetes Mellitus or thyroid dysfunction or cardiac disease. Patients with Thrombocytopenia (<100000/ml), bleeding tendencies, ectopic pregnancy, past history of vascular thrombosis ,uterine anomalies and multiple gestation are excluded from the study.

complete blood picture, urine routine examination, blood sugar, blood grouping, Bleeding Time, Clotting Time, Prothrombin Time, Activated Partial Thromboplastin Time, Hepatitis B Surface Ag, Hepatitis C Virus screening are offered to all patients and findings noted as soon as they conceived. All patients are given routine Folic Acid, Iron and Calcium supplementation orally daily during antenatal period (whether conceived spontaneously or with treatment

200 selected patients with previous unexplained recurrent pregnancy loss are divided into 2 groups:Group A (n = 100) are put on Inj. UFH (Cal-heparin) 5000 U subcutaneous twice daily plus Aspirin 81 mg/day (Juspirin) with the ﬁrst positive pregnancy test, Inj. UFH is given either into anterior abdominal wall or anterior aspect of thigh subcutaneously. While group B (n = 100) receive no thing

ELIGIBILITY:
Inclusion Criteria:

* patients with unexplained recurrent pregnancy loss (RPL)

Exclusion Criteria:

* previous history of Diabetes Mellitus or thyroid dysfunction or cardiac disease
* Thrombocytopenia (<100000/ml)
* bleeding tendencies
* ectopic pregnancy
* past history of vascular thrombosis
* uterine anomalies
* multiple gestation

Ages: 21 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-06-23 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
pregnancy loss | during first 20 weeks of gregnancy
  evidence of abortion is assessed clinically by vaginal bleeding and passage of contents of conception through vagina or by ultrasound through detecting missed abortion .

SECONDARY OUTCOMES:
Maternal outcomes | during 40 weeks of pregnancy
  Maternal outcomes include thromboembolic and hemorrhagic complications and pregnancy-induced hypertension.these outcomes is assessed clinically by follow up mother throughout pregnancy e.g frequent blood pressure monitoring
prematurity | after 20 weeks and before 37 weeks gestation
  delivery of babies before fetal maturity which necessitate admission to the neonatal unit
fetal outcome | during last half of pregnancy(last 20 weeks)
  Foetal growth is monitored by fundal height measurement and serial ultrasounds. Doppler umbilical wave flow velocity is studied for foetuses with suspected intrauterine growth retardation

CONTACTS AND LOCATIONS:
Overall Officials: khalid mohamed, Study Chair — Department of Obstetrics and Gynecology, Benha University Hospital; ahmed saad, Principal Investigator — Benha University; Ibrahim ali, MD, Principal Investigator — Ain Shams University
Locations (1):
- Benha univesity hospital, Banhā, El Qualyobia, Egypt

REFERENCES:
- [Derived] Hamulyak EN, Scheres LJ, Marijnen MC, Goddijn M, Middeldorp S. Aspirin or heparin or both for improving pregnancy outcomes in women with persistent antiphospholipid antibodies and recurrent pregnancy loss. Cochrane Database Syst Rev. 2020 May 2;5(5):CD012852. doi: 10.1002/14651858.CD012852.pub2. PMID 32358837